CLINICAL TRIAL: NCT02020798
Title: Glycemic Response Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Collaborators: Glycemic Index Laboratories, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PEP-1328
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Glycemic Response
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Nutrient formulations without active ingredient (Placebo Comparator): 4 nutrient formulations without active ingredient and variable level of available placebo ingredient
- Nutrient formulation with active ingredien (Experimental): 4 nutrient formulations with increasing amount of active ingredient
  Interventions: Other: Dietary Intervention

INTERVENTIONS:
Other: Dietary Intervention
  Arms: Nutrient formulation with active ingredien

SUMMARY:
The purpose of this study is to assess whether food ingredient(s) affect glycemic responses.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18-75 years of age
* Subject has a body mass index (BMI) ≥ 20.0 and < 35 kg/m² at screening (visit 1).
* Subject has normal fasting serum glucose (<7.0mmol/L capillary corresponding to whole blood glucose <6.3mmol/L).
* Subject has no health conditions that would prevent him from fulfilling the study requirements as judged by the Investigator on the basis of medical history.
* Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study investigator.

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Incremental area under the blood glucose response curve | 0-2 hours
  Glycemic response calculated from individual glucose measurements upon consumption of control and experimental test food products. The individual glucose measurements will be collected at baseline (prior to consumption of each test food product) and over a 2-hour period following the initiation of consumption of each test food product. The primary outcome is differential treatment-effect on the time-concentration glucose curve over the 2 hours post consumption of each test food product.

SECONDARY OUTCOMES:
Rate of decline in blood glucose, peak blood glucose, peak insulin and adjusted time concentration area for insulin | 0-2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto, Canada